CLINICAL TRIAL: NCT03340467
Title: Evaluation of Different Types of Adhesive Materials for Continuous Glucose Monitoring Systems in Subjects With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Adhesive Materials for Continuous Glucose Monitoring Systems
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Metronom Health (Industry)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ADHERE_01
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CGM patch (Experimental): Patient receives four models of CGM patches. Adhesion sites are randomly allocated (1 on each upper arm, 2 on the abdomen).
  Interventions: Device: CGM patch

INTERVENTIONS:
Device: CGM patch — Patient receives four CGM patches.

SUMMARY:
Within the present study 4 different band-aid/adhesive combinations will be tested in patients with type 1 diabetes and type 2 diabetes with regard to adherence to the body and allergic potential. The study period is set to 21 days following adhesive material placement to cover the maximum expected wear-time of the novel CGM system (14 days) plus an additional seven days to ensure that adhesive material is tested for a sufficient time-period and differences in adhesion can clearly be observed.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged ≥18 years
* Type 1 diabetes for at least 6 months according to the WHO definition or Type 2 diabetes for at least 6 months according to the WHO definition
* Body Mass Index (BMI) <45 kg/m²
* Willing and able to wear 4 different band-aid/adhesive materials for the duration of the study and undergo all study procedures
* HbA1c ≤86 mmol/mol

Exclusion Criteria:

* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject
* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods
* Any mental condition rendering the subject incapable of giving his consent
* Subject is using any medication that significantly impacts immune response (oral steroids)
* Has severe medical or psychological condition(s) or chronic conditions/infections that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study
* Subject is actively enrolled in another clinical trial
* Known severe hypersensitivity to adhesive or skin lesions that hinder band-aid application
* Inability of the subject to comply with all study procedures
* Inability of the subject to understand the subject information
* Has children two years of age or younger
* Vulnerable patients, patients deprived from liberty and patients with a physical or mental state altered by disease, age or disability which impacts their ability to defend their interests and for which protection measures are taken ("protected majors" as per French law).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 21 days
  14 days survival rate of different models of CGM patches to fixate a CGM sensor system.

SECONDARY OUTCOMES:
Survival time | 21 days
  Survival time (time to peel-off) of different models of CGM patches to fixate a CGM sensor system
Attachment site reactions | 21 days
  Erythema, edema and blister formation according to ICDRG scoring system

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mader,, Ass Prof, Principal Investigator — Medical University of Graz

IPD SHARING:
Plan to Share IPD: No